CLINICAL TRIAL: NCT06628908
Title: A Phase 3, Randomized, Double-blind, Placebo- and Active-Controlled Study of the Efficacy and Safety of Suzetrigine in Subjects With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Evaluation of Efficacy and Safety of Suzetrigine for Pain Associated With Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-548-110
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Suzetrigine (SUZ) (Experimental): Participants will be randomized to receive SUZ.
  Interventions: Drug: Suzetrigine; Drug: Placebo (matched to Pregabalin)
- Pregabalin (Active Comparator): Participants will be randomized to receive Pregabalin.
  Interventions: Drug: Placebo (matched to SUZ); Drug: Pregabalin
- Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to SUZ and Pregabalin.
  Interventions: Drug: Placebo (matched to SUZ); Drug: Placebo (matched to Pregabalin)

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration.
  Other Names: VX-548; SUZ
  Arms: Suzetrigine (SUZ)
Drug: Placebo (matched to SUZ) — Placebo matched to SUZ for oral administration.
  Arms: Placebo; Pregabalin
Drug: Pregabalin — Capsules for oral administration.
  Arms: Pregabalin
Drug: Placebo (matched to Pregabalin) — Placebo matched to Pregabalin for oral administration.
  Arms: Placebo; Suzetrigine (SUZ)

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of Suzetrigine (SUZ) in participants with pain associated with diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight greater than or equal to (≥) 45 kilogram (kg)
* Body mass index (BMI) ≥18.0 to less than (<) 40.0 kilogram per meter square (kg/m^2)
* Diagnosis of diabetes mellitus type 1 or type 2 by glycosylated hemoglobin A1c (HbA1c) ≤9% and the presence of bilateral pain in lower extremities due to DPN
* Weekly average of daily NPRS score ≥4 and less than or equal to (≤) 9 with limited variation in the 7-day Baseline Period

Key Exclusion Criteria:

* More than 3 missing daily NPRS scores during the 7-day Baseline Period
* Any sensory abnormality (excluding DPN) as pre-specified in the protocol

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Weekly Average of Daily Pain Intensity on the Numeric Pain Rating Scale (NPRS) at Week 12 Compared to Placebo | From Baseline up to Week 12

SECONDARY OUTCOMES:
Change From Baseline in the Medical Outcomes Study 36-item Short-form Health Status (SF 36v2) Physical Component Summary (PCS) Score at Week 12 Compared to Placebo (pooled with data from Study VX24-548-111) | From Baseline up to Week 12
Change From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS at Week 12 Compared to Pregabalin | From Baseline up to Week 12

CONTACTS AND LOCATIONS:
Locations (76):
- United States (76):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Synexus Clinical Research - Birmingham, Birmingham, Alabama
  - AMR Daphne, AL, Daphne, Alabama
  - Synexus Clinical Research - Phoenix Central, Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - Long Beach Research Institute, Long Beach, California
  - Angel City Research, Inc, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - Clinical Trials Research, Sacramento, California
  - Velocity Clinical Research, San Bernardino, San Bernardino, California
  - SCLA Management - Pain Management and Injury Relief, Thousand Oaks, California
  - Diablo Clinical Research (DCR), Walnut Creek, California
  - Velocity Clinical Research - Denver, Englewood, Colorado
  - Velocity Clinical Research - Washington DC, Washington D.C., District of Columbia
  - Accel Research - Deland, DeLand, Florida
  - AMR-Miami, Doral, Florida
  - AMR Fort Myers (The Clinical Study Center), Fort Myers, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - CNS Healthcare - Jacksonville, Jacksonville, Florida
  - Accel Research - St. Petersburg-Largo, Largo, Florida
  - Accel Research - Maitland, Maitland, Florida
  - Suncoast Research Associates - Miami, Miami, Florida
  - 3Sync Research - Miami Lakes, Miami Lakes, Florida
  - Suncoast Clinical Research - New Port Richey, New Port Richey, Florida
  - Synexus Clinical Research - Orlando, Orlando, Florida
  - Conquest Clinical Research - Orlando - Neuro, Orlando, Florida
  - Conquest Clinical Research - Winter Park, Winter Park, Florida
  - Accel Research - Decatur, Decatur, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Feinberg School of Medicine - Anesthesiology, Chicago, Illinois
  - Healthcare Research Network - Flossmoor IL, Flossmoor, Illinois
  - Synexus Clinical Research - Evansville, Evansville, Indiana
  - AMR Wichita East, KS (Heartland Research Associates), Wichita, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Velocity Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research- Covington, Covington, Louisiana
  - Mass General Brigham - Brigham and Women's Hospital - Main Campus, Boston, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Healthcare Research Network - Hazelwood MO, Hazelwood, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - St. Louis Children's Hospital - Nephrology, St Louis, Missouri
  - Synexus Clinical Research - St. Louis, St Louis, Missouri
  - Velocity Clinical Research - Norfolk, Norfolk, Nebraska
  - Synexus Clinical Research - Las Vegas, Las Vegas, Nevada
  - HRI - Hassman Research Institute, Marlton, New Jersey
  - Velocity Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Swift Clinical OpCo, Inc, Brooklyn, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - Synexus Clinical Research - New York (DRS), New York, New York
  - Columbia Presbyterian - The Neurological Institute of New York, New York, New York
  - West Clinical Research, Morehead City, North Carolina
  - Eximia Research - Raleigh, Raleigh, North Carolina
  - Carolinas Pain Institute - Winston-Salem Office, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Synexus Clinical Research - Cincinnati, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Suburban Research Associates - Media, Media, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Synexus Clinical Research- Anderson, Anderson, South Carolina
  - Clinical Trials of South Carolina - Berkeley - Charleston, Charleston, South Carolina
  - M3 Wake Research - Charleston, Charleston, South Carolina
  - Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - AMR Nashville, TN, Nashville, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Synexus Clinical Research - Dallas (DFW) (DRS), Dallas, Texas
  - Be Well Clinical Studies - Austin, Round Rock, Texas
  - San Antonio Clinical Trials, San Antonio, Texas
  - Velocity Clinical Research - Waco, Waco, Texas
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Kalo Clinical Research - West Valley City, West Valley City, Utah
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Northwest Clinical Research Center (NWCRC), Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/